CLINICAL TRIAL: NCT06286319
Title: A Single Center Pilot Study for Cold Oxygen Lung Preservation and Ventilation With the "Angel Cooler"
Brief Title: Cold Oxygen Lung Preservation and Ventilation With the "Angel Cooler"
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: More work needed to modify the device. In addition, more basic animal research needed.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23-00726
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Explanted Lungs (Experimental): After the lungs are explanted from the recipient donor, they will be connected to the "Angel Cooler" via a tracheostomy tube or special adaptor to assess the function of this device in providing cooling oxygen and positive pressure to keep the lungs inflated while on the back table. The lungs will be hooked up to the cooling machine for 15-20 minutes. During this time, investigators will monitor the airway temperature, pressure and oxygen concentration continuously during the entire preservation time. Once these measures are obtained and synced to a corresponding computer, investigators will then disconnect the lungs from the device and continue the standard procedure of sending them to pathology where they will be discarded per usual in lung transplantation.
  Interventions: Device: Angel Cooler

INTERVENTIONS:
Device: Angel Cooler — Device that provides cooled oxygen (between 4-8°C) directly to the lung airways along with external cooling to lung surfaces using cold preservation solutions.

SUMMARY:
The objective of this feasibility study is to evaluate continuous temperature monitoring, oxygen (O2) concentration and ventilation with positive end expiratory pressure (PEEP) to keep lungs cooled at 4-8 degrees Celsius, with continuous O2 concentration of 100% and inflated with a PEEP of 8-10 during the entire cold ischemic period.

DETAILED DESCRIPTION:
The Angel Lung Cooler is a lung preservation method for transplantation. The device has temperature and airway pressure sensors that assess the oxygen temperature in the airways to confirm during the entire preservation time that desired airway temperatures (between 8 and 10 oC) and mean airway pressure to keep the lungs inflated during transportation is optimized.

For the purposes of the trial, the Angel Cooler will be in the operating room at time of transplant when both of the lungs are explanted. The explanted lungs (those removed and not the donor lungs) will be connected to the cooler to determine inflation and temperature changes of the lungs. This procedure will take approximately 5 - 20 minutes. The lungs will then be disconnected from the cooler and then returned to the back table for transport to the Pathology department. As part of standard procedures, the lungs remain in the Operating room for a few hours before they are transported to the Pathology department.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Subjects who have signed Universal Consent are eligible for participation.
* Subjects willing to sign the Universal Consent for the use of their lungs in this study.

Exclusion Criteria:

• Explanted lungs of those who have not signed the Universal Consent (UC) or who have declined participation in the UC will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of Devices Deemed "Functional" | Day 1
  The main outcome is a description of the function of the device (functional/non-functional).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angel, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Study team does not plan to share IPD.